CLINICAL TRIAL: NCT05077735
Title: Stereotactic Biopsy Split-Course Radiation Therapy - Diffuse Midline Glioma (SPORT-DMG)
Brief Title: Stereotactic Biopsy Split-Course Radiation Therapy in Diffuse Midline Glioma, SPORT-DMG Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMROR2162; NCI-2021-10010 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-000069 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Diffuse Midline Glioma, H3 K27M-Mutant
Keywords: DIPG; H3K27M; DMG; Diffuse Midline Glioma
MeSH Terms: interventions — Radiation Dose Hypofractionation; Radiation; Magnetic Resonance Spectroscopy; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (hypofractionated RT) (Experimental): Patients undergo hypofractionated RT over 10 fractions. Patients who achieve progression undergo up to 2 retreatment courses. Patients undergo MRI and PET-CT scan throughout the study.
  Interventions: Radiation: Hypofractionated Radiation Therapy; Other: Questionnaire Administration; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography and Computed Tomography Scan

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated radiation therapy
  Other Names: Hypofractionated; Hypofractionated Radiotherapy; hypofractionation; Radiation, Hypofractionated
Other: Questionnaire Administration — Ancillary studies
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging; Magnetic Resonance / Nuclear Magnetic Resonance; MR; MRI; MR Imaging; MRI Scan; MRIs; NMR Imaging; NMRI; nuclear magnetic resonance imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography and Computed Tomography Scan — Undergo PET-CT scan
  Other Names: PET-CT Scan; PET/CT SCAN; Positron Emission Tomography/Computed Tomography

SUMMARY:
This phase II trial studies the clinical outcomes of hypofractionated radiation therapy in patients with diffuse midline gliomas. This study aims to change the way radiation is delivered, from giving 6 weeks of radiation all at once to giving 2 weeks of radiation. This may determine if there is a difference in the outcome of the treatment, and most importantly, the patients' quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine that 10-month overall survival (OS) rate for the hypofractionated radiation course of 25 Gy in 10 fractions in patients with diffuse midline glioma of the pons isn't inferior to the historical control (survival rate of 50% at 10 months) based on the current standard of care (54 GY in 30 fractions).

SECONDARY OBJECTIVES:

I. To evaluate the quality of life outcomes for patients with diffuse midline gliomas of the pons.

II. To estimate the time to progression after the second hypofractionated radiation course of 25 Gy in 10 fractions in patients with diffuse midline glioma of the pons, calculated from date of diagnosis.

III. To estimate progression free survival intervals for patients after each hypofractionated radiation treatment course.

IV. To evaluate the quality of life outcomes for parents of patients =< 18 years with the Functional Assessment of Cancer Therapy General (FACT-G) Family/Caregiver Questionnaire.

V. To estimate the overall survival for patients with diffuse midline gliomas of the pons treated with planned multi-course hypofractionated radiation courses.

VI. To report toxicities associated with hypofractionated, planned, multi-course radiation treatment for diffuse midline glioma of the pons.

OUTLINE:

Patients undergo hypofractionated radiation therapy (RT) over 10 fractions. Patients who experience progression undergo up to 2 retreatment courses. Patients undergo magnetic resonance imaging (MRI) and positron emission tomography- computed tomography (PET-CT) scan throughout the study.

After completion of study treatment, patients are followed up at 1 month, every 2 months for year 1, every 3 months for year 2, then every 6 months for year 3.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 1 year(s) old (no maximum age)
* Radiologic appearance of diffuse midline glioma of the pons, including diffuse infiltration of >= 50% of the pons on MRI, with or without extension to the midbrain and/or medulla oblongata with at least 1 of the 3 brainstem symptoms (cranial nerve deficit, long tract sign, or cerebellar sign)

  * If all features of this clinicoradiologic criteria are met, then patients can continue on protocol with or without a biopsy
  * If all features of this clinicoradiologic criteria are not met, patients must receive a brainstem lesion biopsy to be treated on protocol. If this cannot be completed, patients will be withdrawn from the study
  * If biopsy has already been completed at an outside institution, the outside pathology report will be reviewed ahead of trial enrollment. The pathology specimen will then be sent to Mayo Clinic for further review, but will not delay study enrollment
* Able to undergo MRI Brain
* Negative urine pregnancy test completed =< 7 days prior to registration, for women of childbearing potential only
* Primary language of English or Spanish for patients and their caregiver
* Patient or caregiver willing and able to provide written informed consent
* Caregiver able to complete questionnaires by themselves or with assistance
* Willing to return to enrolling institution for follow-up during the active monitoring phase of the study

Exclusion Criteria:

* Any patient who has received previous radiation to the brain
* Any patient who has received previous chemotherapy
* Any patient with a diagnosis of neurofibromatosis type 1 or 2 (NF1 or NF2)
* Any of the following:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Other active malignancy =< 5 years prior to registration. EXCEPTIONS: Non-melanotic skin cancer, breast cancer, prostate cancer, well-differentiated thyroid cancer, carcinoma-in-situ of the cervix

  * NOTE: If there is a history or prior malignancy, they must not be receiving other specific treatment for their cancer
* Patients > 16 years with an Eastern Cooperative Oncology Group (ECOG) score >= 4 and patients =< 16 years with a Lansky play scale =< 20

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2027-10-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Time to progression | From date of diagnosis to the date of radiographic or clinical progression following second course of hypofractionated radiation therapy, assessed up to 3 years
  The Wilcoxon Signed-Rank Tests for Non-Inferiority was utilized from PASS software for this design.

SECONDARY OUTCOMES:
Quality of Life Measurement - PedsQL (children under 18) | Baseline up to 3 years
  Results from Pediatric Quality of Life Inventory (PedsQL) Brain Tumor Module will be used to evaluate the quality of life outcomes in patients up to 18 years old. PedsQL™ assessments include 23 items answered on aLikert response scale (0=never a problem; 1=almost never a problem; 2=sometimes a problem; 3=often a problem; 4=almost always a problem) for each item.
Quality of Life Measurement - NFBrSI-24 | Baseline up to 3 years
  The National Comprehensive Cancer Network (NCCN)-Functional Assessment of Cancer Therapy (FACT)-Brain Symptom Index-24 (NFBrSI-24) will be used in patients more than 18 years old. Changes in raw score from baseline to each time-point will be assessed in each of the physical and mental health domains. The NFBrSI-24 consists of 24 questions assessing symptoms over the past 7 days. Items are scored on a 5-point Likert type scale (0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; 4=very much).
Progression free survival | Up to 3 years
  The average progression free survival interval after each course of RT will be reported in months. Progression free survival is defined as the time from registration date to the earliest date of documentation of progression after each course of radiation therapy (RT) or death due to any cause.
FACT-General Family/Caregiver Questionnaire (FACT-G) | Up to 3 years
  Changes in raw score from baseline to each time-point will be assessed in each of the physical and mental health domains. The FACT-G contains 27 questions within 4 subscale domains [Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being] related to health-related quality of life (QOL) in the past 7 days, with higher scoring indicating better QOL.
Overall survival | Up to 3 years
  Overall survival is defined as the time from registration date to death due to any cause. Patients alive at the date of last contact will be censored.
Incidence of adverse events | Up to 3 years
  The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.

CONTACTS AND LOCATIONS:
Overall Officials: Roman O. Kowalchuk, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (2):
- United States (2):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials